CLINICAL TRIAL: NCT00109954
Title: A Prospectively Randomized Controlled Clinical Trial Comparing TheraSphere With Cisplatin-Based TACE (Trans Arterial Chemo Embolization) in the Management of Advanced Stage, Unresectable Hepatocellular Carcinoma (HCC)
Brief Title: Hepatic Arterial Chemoembolization With Cisplatin or Internal Radiation Therapy in Treating Patients With Advanced Liver Cancer That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Weijing Sun, MD, FACP, Professor, University of Pittsburgh
Allocation: Randomized | Purpose: Treatment
Other Study IDs: PCI-04128; CDR0000425333 (Registry Identifier: PDQ (Physician Data Query)); PCI-IRB-0501021
Record Dates: First submitted 2005-05-03; First posted 2005-05-04 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2015-03

CONDITIONS: Liver Cancer
Keywords: adult primary hepatocellular carcinoma; advanced adult primary liver cancer; localized unresectable adult primary liver cancer; recurrent adult primary liver cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Cisplatin; Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: cisplatin
Radiation: brachytherapy
Radiation: yttrium Y 90 glass microspheres

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. In this case, chemotherapy is given through the artery (hepatic artery) that brings blood to the tumor. Chemoembolization kills tumor cells by blocking the blood flow to the tumor and keeping chemotherapy drugs near the tumor. Internal radiation uses radioactive material placed directly into or near a tumor to kill tumor cells. It is not yet known whether hepatic arterial chemoembolization with cisplatin is more effective than internal radiation therapy in treating liver cancer.

PURPOSE: This randomized phase III trial is studying hepatic arterial chemoembolization with cisplatin to see how well it works compared to internal radiation therapy in treating patients with advanced liver cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare time to disease progression in patients with unresectable advanced hepatocellular carcinoma treated with cisplatin-based trans-arterial chemoembolization vs hepatic intra-arterial yttrium Y 90 glass microspheres (TheraSphere®).
* Compare the health-related quality of life of patients treated with these regimens.
* Compare the safety of these regimens in these patients.

Secondary

* Compare survival of patients treated with these regimens.
* Compare tumor response by CT scan in patients treated with these regimens.
* Compare treatment-related costs, in terms of cost of therapy and number of hospitalization days, in these patients.

OUTLINE: This is a randomized study. Patients are stratified according to extent of tumor in the liver (< 50% vs ≥ 50%) and presence of portal hypertension (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo trans-arterial chemoembolization comprising intra-arterial (IA) infusion of cisplatin over 30-60 minutes followed by embolization of the hepatic artery (that brings blood to the tumor) on day 1. Treatment repeats every 8-10 weeks in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive yttrium Y 90 glass microspheres (TheraSphere®) IA on day 1. Beginning 60 days after the first TheraSphere® treatment, patients may receive additional treatment with TheraSphere® only if follow-up CT scans show progressive disease.

Quality of life is assessed at baseline and then every 3 months thereafter.

After the completion of study treatment, patients are followed at 30 days and then every 2 months for 2 years.

PROJECTED ACCRUAL: A total of 120 patients (60 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * Histologically or cytologically confirmed hepatocellular carcinoma (HCC)

    * Confined to the liver
  * Vascular liver mass in the presence of cirrhosis

    * Alpha-fetoprotein level > 500 ng/mL
* Measurable disease

  * At least 1 unidimensionally measurable lesion > 20 mm by spiral CT scan
* Unresectable disease, due to tumor size or extent or presence of cirrhosis
* No metastatic disease, including brain metastases

  * Locoregional lymph node metastases allowed
* No evidence of potential delivery of > 16.5 miCi (30 Gy absorbed dose) of radiotherapy to the lungs either during the first administration of yttrium Y 90 glass microspheres (TheraSphere®) or on cumulative delivery of radiation to the lungs over multiple treatments*
* No evidence of detectable technetium Tc 99m macroaggregated albumin (Tc-99m MAA) flow to the stomach or duodenum after application of established angiographic techniques to stop the flow* NOTE: *For patients randomized to the TheraSphere® arm only

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* More than 12 weeks

Hematopoietic

* WBC > 2,500/mm^3
* Absolute neutrophil count > 1,500/mm^3
* Platelet count > 60,000/mm^3
* No bleeding diathesis not correctable by usual forms of therapy

Hepatic

* See Disease Characteristics
* Bilirubin < 2.0 mg/dL
* AST and/or ALT ≤ 5 times upper limit of normal
* Hepatitis allowed
* No portal hypertension with hepatofugal flow

Renal

* Creatinine < 2.5 mg/dL

Cardiovascular

* No symptomatic congestive heart failure
* No severe peripheral vascular disease that would preclude catheterization

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double barrier or hormonal contraception during and for at least 30 days after completion of study treatment
* No ongoing or active infection
* No other uncontrolled illness
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No more than 1 prior systemic chemotherapy for HCC
* More than 4 weeks since prior IV chemotherapy and recovered
* More than 1 year since prior hepatic arterial cisplatin
* More than 4 months since other prior hepatic arterial chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior external hepatic radiotherapy for HCC

Surgery

* Not specified

Other

* No other concurrent therapy for HCC
* No other concurrent investigational agents

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2005-02; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Progression-free survival as assessed by tumor progression in the treated lobe of the liver
Health-related quality of life at baseline and every 3 months
Toxicity as measured by NCI CTCAE version 3.0

CONTACTS AND LOCATIONS:
Overall Officials: Brian I. Carr, MD, Study Chair — University of Pittsburgh
Locations (1):
- Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania, United States